CLINICAL TRIAL: NCT00551681
Title: Effects of Left Ventricular Pacing Optimilization on Cardiac Perfusion, Contractile Force, and Clinical Performance in Patients With Ventricular Dysfunction and Heart Failure
Acronym: CONTRACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R&D Cardiologie (Other)
Responsible Party: Principal Investigator, Vincent van Dijk, MD, R&D Cardiologie
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDC-2006-04
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Left Ventricular Dysfunction; Heart Failure
Keywords: cardiac resynchronisation therapy; epicardial lead; coronary sinus
MeSH Terms: conditions — Ventricular Dysfunction, Left; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Epicardial left ventricular lead placement
  Interventions: Device: biventricular pacemaker with epicardial left ventricular lead
- 2 (Active Comparator): transvenous left ventricular lead
  Interventions: Device: transvenous left ventricular lead placement

INTERVENTIONS:
Device: biventricular pacemaker with epicardial left ventricular lead — epicardial left ventricular lead placement
  Arms: 1
Device: transvenous left ventricular lead placement — implantation of biventricular pacemaker with transvenous left ventricular lead placement
  Arms: 2

SUMMARY:
To compare a surgical approach of LV lead placement for BIV pacing with the conventional transvenous approach by assessment of differences on the effects on cardiac perfusion and relate this to the clinical cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure NYHA III or IV
* QRS duration >120msec or, when paced > 200msec on 12-lead ECG
* LBBB on ecg
* LV ejection fraction 35% or less
* LV dyssynchony on echocardiography

Exclusion Criteria:

* Severe (drug refractory) heart failure with short (<6 months) life expectancy.
* Permanent or persistent atrial fibrillation
* Other indications for cardiac surgery within 6 months
* Life expectancy less than one year due to other conditions
* Major contra-indication for general anaesthesia
* Participation in another study
* Pregnancy or the desire to become pregnant during the follow up of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-11; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Degree of change in cardiac perfusion following epicardial LV lead placement, compared to transvenous LV lead placement | 6 months

SECONDARY OUTCOMES:
Resynchronization of the LV, measured with TDI, 2D- and 3D-echocardiography, in patients with epicardial LV lead placement, compared to transvenous LV lead placement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lucas VA Boersma, MD, PHD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands